CLINICAL TRIAL: NCT02222831
Title: Optimizing IVF Treatment - the Impact of Time-lapse Culture and Preimplantation Factor (PIF) on Embryo Development.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Regionshospitalet Viborg, Skive (Other)
Responsible Party: Principal Investigator, Betina Boel Povlsen, MSc, MSc, Laboratory Director, The Fertility Clinic Skive; Denmark., Regionshospitalet Viborg, Skive
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Skive-2014-BBP
Record Dates: First submitted 2014-08-20; First posted 2014-08-21 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: In Vitro Fertilization; Assisted Reproductive Techniques
Keywords: IVF; Embryo Quality; Time Lapse Culture; Preimplantation factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Day 0 - Study arm (Experimental): Day 0 denudation and time lapse culture on IVF-oocytes.:
  After insemination the oocytes will subsequently be denuded and cultured in the EmbryoScope (day 0).
  The embryo culture media will be collected at day 2-5.
  Interventions: Procedure: Day 0 denudation and time lapse culture on IVF-oocytes.
- Day 1 - control arm (No Intervention): After insemination oocytes in the control group will be incubated in a standard incubator overnight. On day 1 the oocytes in the will be denuded and further cultured in the EmbryoScope.
  The embryo culture media will be collected at day 2-5.

INTERVENTIONS:
Procedure: Day 0 denudation and time lapse culture on IVF-oocytes.
  Arms: Day 0 - Study arm

SUMMARY:
The aims of this study are to evaluate:

1. the possible effect of time-lapse culture from day zero (day of oocyte retrieval) on fertilisation rates and embryo quality in standard IVF.
2. the association between PIF status in embryo culture medium and embryo quality assessed by standard subjective parameters and morphokinetic development.

ELIGIBILITY:
Inclusion Criteria:

* Standard IVF treatment
* Body mass Index (BMI) between 18 and 30
* couples in which the male partner has normal sperm concentration and motility according to the World Health Organization (WHO, 2010)

Exclusion Criteria:

- Patients with less than four oocytes

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-01 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Embryo Quality | Day 0-5 after oocyte pick-up

SECONDARY OUTCOMES:
Fertilisation rate | Day 1 after oocyte pick-up

OTHER OUTCOMES:
Clinical pregnancy rate | 7th week of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Betina B Povlsen, MSc, Principal Investigator — The Fertility Clinic, Skive Regional Hospital, Denmark
Locations (1):
- The Fertility Clinic Skive, Skive, Denmark